CLINICAL TRIAL: NCT04741087
Title: A Combined Phase 2/3 12-week, Randomized, Double-blind, Placebo-controlled Study Investigating the Efficacy of AMT-101 in Subjects With Chronic Antibiotic-resistant Pouchitis
Brief Title: Study of the Safety and Efficacy of AMT-101 in Subjects With Pouchitis
Acronym: FILLMORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Applied Molecular Transport (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMT-101-201
Record Dates: First submitted 2021-01-15; First posted 2021-02-05 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-04

CONDITIONS: Pouchitis
Keywords: Inflammatory Bowel Disease
MeSH Terms: conditions — Pouchitis; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMT-101 (Dose A) (Active Comparator): Dose A: AMT-101 Tablet
  Interventions: Drug: AMT-101 (oral)-Dose A
- AMT-101 (Dose B) (Active Comparator): Dose B: AMT-101 Tablet
  Interventions: Drug: AMT-101 (oral)-Dose B

INTERVENTIONS:
Drug: AMT-101 (oral)-Dose A — AMT-101 is an orally administered biologic therapeutic, taken once daily.
  Arms: AMT-101 (Dose A)
Drug: AMT-101 (oral)-Dose B — AMT-101 is an orally administered biologic therapeutic, taken once daily.
  Arms: AMT-101 (Dose B)

SUMMARY:
Phase 2 Study Investigating the Efficacy of AMT-101 in Subjects with Chronic Antibiotic-resistant Pouchitis

DETAILED DESCRIPTION:
A Phase 2 12-week, Randomized, Double-blind, Placebo-controlled Study Investigating the Efficacy of AMT-101 in Subjects with Chronic Antibiotic-resistant Pouchitis

ELIGIBILITY:
Inclusion Criteria:

• Chronic or recurrent pouchitis

Exclusion Criteria:

* Known gastrologic, or systemic condition that may compromise severity or diagnosis of disease.
* History or current evidence of colonic or abdominal abnormalities.
* Previous exposure to AMT-101 or similar and known hypersensitivity to AMT-101 or its excipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Stool Frequency Response | 12 weeks
Histologic Healing | 12 weeks
  based upon the Geboes scoring system and PDAI

SECONDARY OUTCOMES:
Histologic Response | 12 weeks
  based upon the Geboes scoring system and PDAI
Change in Endoscopic Score | 12 weeks
Change in Stool Frequency | 12 weeks

CONTACTS AND LOCATIONS:
Locations (34):
- United States (12):
  - Connecticut Clinical Research Institute, Bristol, Connecticut
  - University of Chicago Medical Center, Chicago, Illinois
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Gastrointestinal Associates - Jackson, Flowood, Mississippi
  - University of North Carolina GI, Chapel Hill, North Carolina
  - Gastro One, Germantown, Tennessee
  - Gastrointestinal Asssociates- GIA Clinical Trials, LLC, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Tyler Research Institute, LLC, Tyler, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Washington Gastroenterology, Tacoma, Tacoma, Washington
- Belgium (2):
  - UZ Leuven - University Hospital Gasthuisberg, Leuven
  - Groupe santé CHC / Clinique du MontLégia, Liege, Liège
- GI Research Institute, Vancouver, British Columbia, Canada
- France (4):
  - CHU de Rennes - Hopital de Pontchaillou, Rennes
  - CHU Saint Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
  - CHRU Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (4):
  - Praxis fur Gastroenterologie am Bayerischen Platz, Berlin
  - Klinik für Innere Medizin KIM IV, Jena
  - UKSH Universitätsklinikum Schleswig-Holstein, Kiel
  - University Hospital Tübingen, Tübingen
- Hungary (2):
  - Semmelweis Egyetem I. sz Belgyogyaszati Klinika, Budapest
  - Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar, Szeged
- ETZ - Elisabeth, Tilburg, Netherlands
- Hospital Universitario y Politecnico La Fe de Valencia, Valencia, Spain
- Switzerland (2):
  - Clarunis Bauchzentrum, Basel
  - University Hospital of Zürich, Zurich
- United Kingdom (5):
  - MAC Clinical Research - Blackpool, Blackpool, Lancashire
  - MAC Clinical Research - Liverpool, Prescot, Liverpool
  - MAC Clinical Research - Cannock, Cannock, South Staffordshire
  - MAC Clinical Research - Leeds, Leeds, West Yorkshire
  - MAC Clinical Research - Manchester, Manchester